CLINICAL TRIAL: NCT01149564
Title: Comparison of Oral and Intravenous Ibuprofen for Treatment of Patent Ductus Arteriosus in Extremely Premature Infants: A Randomized Controlled Trial
Brief Title: Comparison of Oral and Intravenous Ibuprofen for PDA Treatment in Premature Infants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chairman of Department of Pediatrics, China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR-99; DMR-98 (Other Grant/Funding Number: China Medical University Hospital)
Record Dates: First submitted 2010-06-20; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Extremely Premature Infants; PDA; Oral Ibuprofen; IV Ibuprofen
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV ibuprofen (Placebo Comparator): The first dose of either oral or IV ibuprofen will be given at the time the patient is randomized.The subsequent doses of indometacin or ibuprofen are also determined according to the echocardiographic PDA flow patterns at intervals of once every 24 hours from the last dose. The dosage of both oral ibuprofen (Ibuprofen suspension, 20 mg/ml, Yung Shing Co., Taiwan) and IV ibuprofen (PedeaR 20 mg/ml, developed by Orphan Europe and approved by the EMEA) are an initial dose of 10 mg/kg and then 5 mg/kg at 24-hour intervals as indicated by PDA flow pattern.
  Interventions: Drug: iv ibuprofen
- Oral ibuprofen (Active Comparator)
  Interventions: Drug: oral ibuprofen

INTERVENTIONS:
Drug: iv ibuprofen
  Arms: IV ibuprofen
Drug: oral ibuprofen
  Arms: Oral ibuprofen

SUMMARY:
Background:

Patent ductus arteriosus (PDA) continues to be one of the most common problems in premature infants. Pharmacological closure of PDA with intravenous (IV) indomethacin was first reported in 1976, however, concern remains regarding the safety of indomethacin, which affects renal, GI and cerebral perfusion and may lead to complications such as transient or permanent renal dysfunction, NEC, GI hemorrhage, and reduced cerebral oxygenation. Recently, IV ibuprofen has been shown to be effective for the closure of patent ductus arteriosus in premature infants, without reducing mesenteric, renal, or cerebral blood flow. We have developed the echocardiographic PDA flow pattern as a guide for PDA treatment, fewer doses of drugs were needed to achieve acceptable closing rates. We have also reported that IV ibuprofen is as effective as IV indometacin for the PDA treatment in extremely premature infants, without increasing the incidence of complications in a randomised controlled trial. Several studies reported that oral ibuprofen may be effective for PDA treatment. To date there is no firm conclusion as to the efficacy and safety of oral ibuprofen compared with IV ibuprofen for PDA closure in extremely premature infants.

Objective:

Since the efficacy of pharmacological closure of PDA is related to gestational age, and extremely premature infants carry the highest rate of mortality and morbidity. We intend to conduct a randomized controlled trial to compare oral and intravenous ibuprofen for treatment of PDA in this high-risk population of extremely premature infants.

Methods:

Extremely premature infants (gestational age < 28 weeks) admit to the NICU will be eligible for enrollment. Informed parental consent will be obtained according to the Institutional Review Board's instructions. Extremely premature infants with respiratory distress syndrome (RDS) and PDA confirmed by echocardiography will be randomly assigned to receive either oral or IV ibuprofen. The subsequent doses of ibuprofen are also determined according to our specific echocardiographic PDA flow patterns at intervals of once every 24 hours from the last dose. The dosage of oral or ibuprofen is 10 mg/kg (1 ml) and then 5 mg/kg at 24-hour intervals as indicated by echocardiographic PDA flow pattern.

Sample Size Calculation and Length of the Study Period:

About 50-60 extremely premature infants will be admitted to our NICU each year. To prove with McNemar's Test at a one-sided significance level of 5% and a power of 90% that using oral ibuprofen instead of IV ibuprofen results in comparable PDA closure rates, only 31 extremely premature infants with RDS and PDA have to be enrolled. Allowing for attrition and exclusion from the final study groups, the length of the study period will be safe to set to 2 years.

Expected Results:

We expect to determine whether oral ibuprofen is effective and safe in inducing PDA closure in extremely premature infants and to compare the complications between infants treated with oral ibuprofen and those with IV ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* premature infants gestational age < 28 weeks, respiratory distress syndrome requiring assisted ventilation, a PDA without other cardiac anomalies confirmed by echocardiography within 24 hours after birth,

Exclusion Criteria:

* severe congenital anomalies or lethal cardiopulmonary conditions, and informed consent could be obtained from parents

Ages: 3 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to ascertain whether oral ibuprofen is effective and safe in inducing PDA closure in extremely premature infants. | 1 month
  Number of extremely premature infants with PDA closed or Adverse Events as a Measure of efficiency and safety.

SECONDARY OUTCOMES:
A secondary objective is to compare the complications between infants treated with oral ibuprofen and those treated with IV ibuprofen. | 1 month
  Number of extremely premature infants in each group with PDA closed or Adverse Events as a Measure of efficiency and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Horng Su, MD, PhD, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan